CLINICAL TRIAL: NCT05907772
Title: Incorporation of Protein Induced by Vitamin K Absence or Antagonist-II Into Transplant Criteria Expands Beneficiaries of Liver Transplantation for Hepatocellular Carcinoma: A Multi-center Retrospective Cohort Study in China
Brief Title: Incorporation of Protein Induced by Vitamin K Absence or Antagonist-II Into Transplant Criteria Expands Beneficiaries of Liver Transplantation for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2023-ZJU-OBS1
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cancer of Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recipients with preoperative PIVKA-II≤240mAU/mL
  Interventions: Other: No intervention
- Recipients with preoperative PIVKA-II>240mAU/mL
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a multi-center study in China to investigate the role of PIVKA-II in HCC recipient selection and prognostic stratification by analyzing the data of 522 recipients with HCC registered in the China Liver Transplant Registry.

ELIGIBILITY:
Inclusion Criteria:

* The HCC patients received LT with pre-operative PIVKA-II records performed from January 2015 to December 2020, whose clinicopathological data were registered in the CLTR.

Exclusion Criteria:

* (1) patients who received split LT or simultaneous transplantation, (2) patients who received re-transplantation, (3) patients with macroscopic portal vein tumor thrombosis or other macrovascular invasion, (4) patients with incomplete follow-up or incomplete important parameters records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 522 HCC patients underwent liver transplant with pre-operative PIVKA-II records were studied.
Sampling Method: Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2022-08-27 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | January 2015 to December 2020
  the overall survival of liver transplant recipient with HCC

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Dong L, Lu Q, Yang Z, Fan X, Gao F, Ge W, Wang Z, Zhou Z, Lu D, Wei X, Wei Q, Zhuang L, Qin L, Ye Q, Yang J, Dong J, Zheng S, Xu X. Incorporation of protein induced by vitamin K absence or antagonist-II into transplant criteria expands beneficiaries of liver transplantation for hepatocellular carcinoma: a multicenter retrospective cohort study in China. Int J Surg. 2023 Dec 1;109(12):4135-4144. doi: 10.1097/JS9.0000000000000729. PMID 37988413